CLINICAL TRIAL: NCT06052202
Title: Reducing Colorectal Cancer Health Disparities: An mHealth Intervention to Improve Screening Among African American Men
Brief Title: A Smartphone-Based Intervention to Improve Colorectal Cancer Screening in African American Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISA Associates, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R44CA246899 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRC mHealth intervention (Experimental): Experimental group participants will have access to the CRC mHealth intervention.
  Interventions: Behavioral: CRC mHealth
- Control Education (Active Comparator): Control condition participants will receive information about colorectal cancer and screening developed by the Centers for Disease Control.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: CRC mHealth — Participants receive text messages that contain information about colorectal cancer and screening. Some text messages include links to videos that are intended to reduce barriers to colorectal cancer screening. Other text messages include links to brief web-based assessments. Responses to assessment questions are used to make sure each man receives only the information relevant to his needs. The main educational content is completed in the first 6 weeks. Additional educational and motivation text messages continue for up to 4 more months if a participant reports not having completed colorectal cancer screening.
  Arms: CRC mHealth intervention
Behavioral: Control — Participants receive text messages that include links to videos and/or brochures developed by the Centers for Disease Control. This information is designed to educate the public about colorectal cancer and motivate screening. Text messages are sent every 2-3 days for 6 weeks.
  Arms: Control Education

SUMMARY:
The goal of this clinical trial is to test a new smartphone-based program designed to help African American men get screened for colorectal cancer (CRC). The main question it aims to answer is:

° Are African American men who complete the smartphone-based program more likely to get screened for colorectal cancer than men who do not?

Participants will:

* Complete a baseline survey asking about their colorectal cancer screening history and their thoughts and beliefs about colorectal cancer and the medical system.
* Be randomized to receive the new smartphone-based program or to receive text messages containing colorectal cancer education materials designed by the Centers for Disease Control (CDC). The new program sends text messages with information about colorectal cancer. Some of these text messages have links to videos that try to help men overcome anything that may stand in the way of getting screened.
* Complete a follow-up survey 6 months after the baseline survey. This survey will ask the same questions as the baseline survey.
* A medical records review will be conducted at 6 months to verify whether participants received a colorectal cancer screening test during the study period.

Researchers will compare participants who receive the new smartphone-based program to participants who receive the CDC information. The goal is to see whether the smartphone-based program increasing screening more than standard educational materials available on the internet.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black
* not compliant with current United States Preventive Services Taskforce colorectal cancer screening recommendations
* owns a mobile phone capable of text messaging and accessing webpages
* able to speak/understand English

Exclusion Criteria:

* personal history of colorectal cancer

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha L Leaf, Ph.D., Principal Investigator — ISA Associates
Locations (1):
- ISA Associates, Inc., Alexandria, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRC mHealth Intervention | Control Education
Started | 63 | 65
Completed | 47 | 47
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRC mHealth Intervention | Control Education | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (7.2) | 56.2 (6.8) | 56.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 63 | 65 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 62 | 123
  White | 0 | 0 | 0
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 63 | 64 | 127
  Unknown or Not Reported | 0 | 0 | 0
Percentage of Participants Reporting Yes to Receiving a Colorectal Cancer Screening Test [Number; unit: percentage of participants screened] — Participants responded to a multiple-choice item asking whether they had ever completed a recommended colorectal cancer screening (colonoscopy, FIT, FIT-DNA, virtual colonoscopy, or flexible sigmoidoscopy). Participants reported lifetime receipt at baseline. Response options were Yes/No/I'm not sure.
  percentage of participants screened | 52.4 | 49.2 | 50.8
Perceived Severity of Colorectal Cancer [Mean (Standard Deviation); unit: units on a scale] — Measured using the 12-item perceived severity subscale of Green and colleagues' (2004) CRC Knowledge, Perceptions, and Screening Survey. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived severity.
  units on a scale | 3.22 (0.75) | 3.03 (0.78) | 3.12 (0.77)
Perceived Susceptibility to Colorectal Cancer [Mean (Standard Deviation); unit: units on a scale] — Measured using the 5-item perceived susceptibility subscale of Green and colleagues' (2004) CRC Knowledge, Perceptions, and Screening Survey. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived susceptibility.
  units on a scale | 2.77 (0.60) | 2.67 (0.83) | 2.72 (0.73)
Perceived Benefits to Colonoscopy [Mean (Standard Deviation); unit: units on a scale] — Measured using Rawl and colleagues' (2001) 5-item perceived benefits to colonoscopy scale. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived benefits to colonoscopy.
  units on a scale | 4.08 (0.53) | 4.03 (0.54) | 4.06 (0.54)
Perceived Benefits to Stool Test [Mean (Standard Deviation); unit: units on a scale] — Measured using Rawl and colleagues' (2001) 5-item perceived benefits to fecal occult blood test scale. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived benefits to stool tests.
  units on a scale | 3.86 (0.51) | 3.95 (0.55) | 3.91 (0.53)
Colorectal Cancer Knowledge [Mean (Standard Deviation); unit: units on a scale] — Measured using the 16-item CRC Knowledge test subsection of Green and colleagues' (2004) CRC Knowledge, Perceptions, and Screening Survey. The true/false items are scored 1 (correct) or 0 (incorrect) and summed to form a score ranging from 0 to 16. Higher scores indicate greater colorectal cancer knowledge.
  units on a scale | 13.33 (1.76) | 13.37 (1.80) | 13.35 (1.77)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Received a Colorectal Cancer Screening Test
Description: This measure assesses whether or not a participant received a colorectal cancer screening test since beginning the study. The date and type of screening will be verified via electronic health records. A value of "0" will be recorded if no screening test is found in the electronic health record. A value of "1" will be recorded if a screening test is found in the electronic health record. The percentage of participants with a electronic health record verified screening will be calculated from these values.
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 63 | 65
Participants | 2 | 2

2. Secondary Outcome: Perceived Severity of Colorectal Cancer at Month 6
Description: Measured using the 12-item perceived severity subscale of Green and colleagues' (2004) CRC Knowledge, Perceptions, and Screening Survey. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived severity.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 47 | 47
units on a scale | 2.82 (0.76) | 2.59 (0.61)

3. Secondary Outcome: Perceived Susceptibility to Colorectal Cancer at Month 6
Description: Measured using the 5-item perceived susceptibility subscale of Green and colleagues' (2004) CRC Knowledge, Perceptions, and Screening Survey. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived susceptibility.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 47 | 47
units on a scale | 2.82 (0.76) | 2.59 (0.61)

4. Secondary Outcome: Perceived Benefits to Colonoscopy at Month 6
Description: Measured using Rawl and colleagues' (2001) 5-item perceived benefits to colonoscopy scale. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived benefits to colonoscopy.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 47 | 47
units on a scale | 4.23 (0.51) | 4.11 (0.54)

5. Secondary Outcome: Perceived Benefits to Stool Test at Month 6
Description: Measured using Rawl and colleagues' (2001) 5-item perceived benefits to fecal occult blood test scale. Items are averaged to form a score ranging from 1 to 5 with higher scores indicating higher perceived benefits to stool tests.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 47 | 47
units on a scale | 3.91 (0.52) | 4.06 (0.52)

6. Secondary Outcome: Colorectal Cancer Knowledge at Month 6
Description: Measured using the 16-item CRC Knowledge test subsection of Green and colleagues' (2004) CRC Knowledge, Perceptions, and Screening Survey. The true/false items are scored 1 (correct) or 0 (incorrect) and summed to form a score ranging from 0 to 16. Higher scores indicate greater colorectal cancer knowledge.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 47 | 47
score on a scale | 13.70 (1.49) | 13.17 (1.43)

7. Primary Outcome: Percentage of Participants Reporting Yes to Receiving a Colorectal Cancer Screening Test
Description: Participants responded to a multiple-choice item asking whether they had completed a recommended colorectal cancer screening (colonoscopy, FIT, FIT-DNA, virtual colonoscopy, or flexible sigmoidoscopy) in the past 6 months. Response options were Yes/No/I'm not sure.
Time Frame: baseline, 6-months
Measure: Number (95% Confidence Interval); unit: Percentage of participants screened
Arm/Group | CRC mHealth Intervention | Control Education
Number analyzed (Participants) | 47 | 47
Percentage of participants screened | 40.4 [27.6 to 54.7] | 17.0 [8.9 to 30.1]

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to approximately 6 months
Arm/Group | CRC mHealth Intervention | Control Education
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/65
Other Adverse Events (participants affected / at risk) | 0/63 | 0/65

LIMITATIONS AND CAVEATS:
The planned primary outcome -EHR-verified CRC screening - could not be assessed due to failed record linkage. The clinic initially confirmed that name and phone number would suffice, but immediately before extraction FMCS required additional identifiers (e.g., date of birth) to match most records. Despite multiple attempts at alternative matching, linkage remained inadequate, leaving the EHR data unusable for the endpoint. We therefore report survey-based proxy composite outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT06052202/Prot_SAP_000.pdf